CLINICAL TRIAL: NCT03523715
Title: Effect of Prunes on Gastrointestinal Function After Gynecological Surgery: A Randomized Controlled Trial
Brief Title: Prunes for Gastrointestinal Function After Gynecologic Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruiting participants
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Begum Ozel, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-17-00548
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Dioctyl Sulfosuccinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prunes (Experimental): The study group will be instructed to consume 4 oz of prunes as well as docusate sodium twice daily for 3 days after surgery.
  Interventions: Dietary Supplement: Prunes; Drug: Docusate Sodium
- Control (Placebo Comparator): The placebo group will be instructed to take docusate sodium twice daily for 3 days after surgery.
  Interventions: Drug: Docusate Sodium

INTERVENTIONS:
Dietary Supplement: Prunes — 12 oz of prunes daily
  Other Names: Dried plums
  Arms: Prunes
Drug: Docusate Sodium — Oral docusate sodium twice daily
  Other Names: Colace

SUMMARY:
This is a prospective, randomized control trial that randomizes patients post-operatively into standard care versus standard care plus prunes. Patients in the control arm will take 100 mg docusate twice per day for 3 days (standard care). Participants in the treatment arm will consume 4 oz prunes daily and take 100 mg docusate twice per day for 3 days. The primary objective is to determine the time to first bowel movement after surgery.

DETAILED DESCRIPTION:
A major postoperative complaint among benign gynecological surgery patients is constipation. Improved management of constipation among these patients has the potential to both alleviate pain and for significant savings for health care systems. This is a prospective, randomized control trial that randomizes patients post-operatively into standard care versus standard care plus prunes. The primary objective is to determine the time to first bowel movement after surgery. Secondary objectives are pain associated with first bowel movement, stool consistency using Bristol stool form scale, compliance and patient satisfaction. The study population includes women over the age of 18 undergoing benign gynecologic surgery with overnight stay. Patients in the control arm will take 100 mg docusate twice per day for 3 days (standard care). Participants in the treatment arm will consume 4 oz prunes daily and take 100 mg docusate twice per day for 3 days. Follow-up phone calls will be made 3 and 5 days postoperatively to inquire about primary and secondary outcomes. Participants will be randomized to the treatment or control group at a 1:1 ratio and using randomization blocks of 6. Participant characteristics will be presented as means and standard deviations for continuous variables and counts and percentages for categorical variables. The primary and secondary outcomes will be assessed using two-sample t-tests.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients seen in the Gynecology or Urogynecology clinics at LAC+USC Medical Center who are planned for surgery requiring at least 24 hour stay
2. Age 18 or greater
3. Able to give informed consent
4. No contraindications to docusate or prune consumption

Exclusion Criteria:

1. Unable to give informed consent
2. Unwilling to follow protocol
3. Active malignancy
4. Emergency surgery
5. Diabetes mellitus
6. Inflammatory bowel disease, gastroparesis, or other bowel disorder
7. History of bowel resection or presence of colostomy
8. Dependence on regular laxative use prior to surgery
9. Baseline frequency of bowel movements less than weekly
10. Intraoperative enterotomy or any bowel surgery performed at the time of surgery
11. Patient unable to initiate oral intake on post op day 1 for any reason
12. Allergy to docusate or prunes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Begum Ozel, MD, Principal Investigator — Keck School of Medicine
Locations (1):
- Los Angeles Count + USC Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel M, Schimpf MO, O'Sullivan DM, LaSala CA. The use of senna with docusate for postoperative constipation after pelvic reconstructive surgery: a randomized, double-blind, placebo-controlled trial. Am J Obstet Gynecol. 2010 May;202(5):479.e1-5. doi: 10.1016/j.ajog.2010.01.003. Epub 2010 Mar 6. PMID 20207340
- [Background] McNanley A, Perevich M, Glantz C, Duecy EE, Flynn MK, Buchsbaum G. Bowel function after minimally invasive urogynecologic surgery: a prospective randomized controlled trial. Female Pelvic Med Reconstr Surg. 2012 Mar-Apr;18(2):82-5. doi: 10.1097/SPV.0b013e3182455529. PMID 22453316
- [Background] Lever E, Cole J, Scott SM, Emery PW, Whelan K. Systematic review: the effect of prunes on gastrointestinal function. Aliment Pharmacol Ther. 2014 Oct;40(7):750-8. doi: 10.1111/apt.12913. Epub 2014 Aug 11. PMID 25109788
- [Background] Lever E, Scott SM, Louis P, Emery PW, Whelan K. The effect of prunes on stool output, gut transit time and gastrointestinal microbiota: A randomised controlled trial. Clin Nutr. 2019 Feb;38(1):165-173. doi: 10.1016/j.clnu.2018.01.003. Epub 2018 Feb 15. PMID 29398337
- [Background] Attaluri A, Donahoe R, Valestin J, Brown K, Rao SS. Randomised clinical trial: dried plums (prunes) vs. psyllium for constipation. Aliment Pharmacol Ther. 2011 Apr;33(7):822-8. doi: 10.1111/j.1365-2036.2011.04594.x. Epub 2011 Feb 15. PMID 21323688
- [Derived] Rasouli MA, Dancz CE, Dahl M, Volpe KA, Horton CJ, Ozel BZ. Effect of prunes on gastrointestinal function after benign gynecological surgery: a randomized control trial. Langenbecks Arch Surg. 2022 Dec;407(8):3803-3810. doi: 10.1007/s00423-022-02584-8. Epub 2022 Jun 22. PMID 35732845

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prunes | Control
Started | 38 | 39
Completed | 26 | 23
Not Completed | 12 | 16
Not completed — Lost to Follow-up | 11 | 14
Not completed — Did not meet inclusion criteria | 1 | 0
Not completed — Internally inconsistent reporting | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prunes | Control | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (9.9) | 51.1 (10.6) | 50 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 20 | 42
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 7 | 14 | 21
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 15 | 9 | 24
Post menopause [Count of Participants; unit: Participants] | 9 | 11 | 20
Baseline Bristol Stool Scale [Median (Inter-Quartile Range); unit: units on a scale] | 4 [3 to 5] | 4 [3 to 4] | 4 [3 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Time to First Bowel Movement
Description: Time to first bowel movement after surgery
Time Frame: 3 days
Measure: Mean (Standard Deviation); unit: hours post surgery
Arm/Group | Prunes | Control
Number analyzed (Participants) | 26 | 24
hours post surgery | 57.6 (19.3) | 53.8 (21.7)

2. Secondary Outcome: Stool Consistency of the First Bowel Movement
Description: Bristol Stool chart in which stool consistency is described as type 1 to 7 with higher values indicating more liquid stool
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: Bristol Stool Scale
Arm/Group | Prunes | Control
Number analyzed (Participants) | 26 | 24
Bristol Stool Scale | 3 [2 to 5] | 4 [2 to 6]

3. Secondary Outcome: Pain With Bowel Movement Measured
Description: Likert scale from 0 to 10 in which higher values indicate more pain
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: Likert scale 0-100
Arm/Group | Prunes | Control
Number analyzed (Participants) | 26 | 24
Likert scale 0-100 | 60 [25 to 80] | 40 [10 to 70]

4. Secondary Outcome: Satisfaction With Bowel Regimen
Description: Likert scale from 0 to 10 in which higher values indicate more satisfaction
Time Frame: 3 day
Measure: Median (Inter-Quartile Range); unit: Likert scale 0-100
Arm/Group | Prunes | Control
Number analyzed (Participants) | 26 | 24
Likert scale 0-100 | 100 [70 to 100] | 80 [45 to 95]

5. Secondary Outcome: Satisfaction With Surgery Overall
Description: Likert scale from 0 to 10 in which higher levels indicate more satisfaction
Time Frame: 3 days
Measure: Median (Inter-Quartile Range); unit: Likert scale 0-100
Arm/Group | Prunes | Control
Number analyzed (Participants) | 26 | 24
Likert scale 0-100 | 100 [90 to 100] | 100 [97.5 to 100]

6. Secondary Outcome: Requirements for Laxatives
Description: The number of participants who used any laxatives (besides the prunes and stool softeners) during the study period.
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prunes | Control
Number analyzed (Participants) | 26 | 24
Participants | 7 | 6

7. Secondary Outcome: Bowel Movement in the Study Period
Description: The number of participants who had a bowel movement in the post operative study follow up
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prunes | Control
Number analyzed (Participants) | 26 | 24
Participants | 26 | 17

ADVERSE EVENTS:
Time Frame: The study follow up period was 5 days.
Arm/Group | Prunes | Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/24
Other Adverse Events (participants affected / at risk) | 0/26 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT03523715/Prot_SAP_ICF_000.pdf